CLINICAL TRIAL: NCT06165393
Title: The Effect of Alginate Encapsulated Supplements on Athletic Performance and Recovery
Acronym: SWAP
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Aarhus (Other)
Collaborators: Innovation Fund Denmark (Individual)
Responsible Party: Principal Investigator, Per Bendix Jeppesen, Associate. Prof, PhD., University of Aarhus
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Other
Other Study IDs: SWAP AU
Record Dates: First submitted 2023-12-01; First posted 2023-12-11 (Actual); Last update posted 2023-12-11 (Actual); Status verified 2023-12

CONDITIONS: Athletic Performance

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Slow-release CHO-AA (Experimental): Alginate encapsulated Carbohydrates and Amino Acids
  Interventions: Dietary Supplement: Slow-release CHO-AA
- Slow-release CHO (Experimental): Alginate encapsulated Carbohydrates
  Interventions: Dietary Supplement: Slow-release CHO
- CHO (Active Comparator): Carbohydrates only
  Interventions: Dietary Supplement: CHO

INTERVENTIONS:
Dietary Supplement: Slow-release CHO-AA — Slow-release CHO-AA, alginate encapsulated
  Arms: Slow-release CHO-AA
Dietary Supplement: Slow-release CHO — Slow-release CHO, alginate encapsulated
  Arms: Slow-release CHO
Dietary Supplement: CHO — Carbohydrate-only, control
  Arms: CHO

SUMMARY:
Endurance sport is often characterized by high training loads and significant metabolic demands, including depletion of endogenous fuel stores (e.g. liver and muscle glycogen) and damage to the skeletal muscle proteins. Nutritional interventions that enhance the restoration of endogenous fuel stores and improve muscle damage repair have received a lot of attention. The primary aim of this project is to clinically test the effect of alginate encapsulation technology on performance. Furthermore, we will investigate the substrate utilization profile during exercise and subsequent recovery.

The encapsulation technology presents a nutrient delivery solution, which results in a sustained or slow-release of the nutrients encapsulated. Thus, potentially optimizing the digestion and absorption by promoting an easy ingestion of high concentrations of fx carbohydrates without negatively affecting the gastrointestinal comfort.

ELIGIBILITY:
Inclusion Criteria:

* males between 18-50 years of age
* moderate to trained individuals with a VO2max > 50 ml/min/kg
* accustumed to exercising on a bike
* healthy volunteers

Exclusion Criteria:

* persons diagnosed with metabolic diseases (i.e. Type 2 Diabetes) which relates to the carbohydrate metabolism.
* persons ingesting prescribed drugs/medicin, supplements or a special diet (i.e. low carbohydrate), which might affect the glycogen synthesis and/or performance.

Ages: 18 Years to 50 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes
Enrollment: 20 (Estimated)
Dates: Start 2022-05-11 (Actual); Primary Completion 2023-12-01 (Estimated); Study Completion 2023-12-31 (Estimated)

PRIMARY OUTCOMES:
Performance | approx. 90 min-120 min
  Time-To-Exhaustion performance test

CONTACTS AND LOCATIONS:
Locations (1):
- Per Bendix Jeppesen, Aarhus N, Denmark